CLINICAL TRIAL: NCT00234702
Title: A Phase II, Double-blind, Randomized, Placebo-controlled Study to Assess the Efficacy and Safety of Lanthanum Carbonate for the Reduction of Serum Phosphorus in Subjects With Stage 3 and 4 Chronic Kidney Disease Who Have Elevated Serum Phosphorus Levels
Brief Title: Efficacy and Safety of Lanthanum Carbonate in Reducing Serum Phosphorus Levels in Subjects With Stage 3 and 4 Chronic Kidney Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPD405-206
Record Dates: First submitted 2005-10-05; First posted 2005-10-07 (Estimated); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Kidney Diseases
MeSH Terms: conditions — Kidney Diseases | interventions — lanthanum carbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Lanthanum carbonate
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lanthanum carbonate — Lanthanum carbonate 750mg/day, T.I.D. for 2 weeks; titrated at the next 3 weekly visits in order to achieve target serum phosphorus levels, up to a maximum dose of 3000mg/day; 4-week maintenance period where subject receives the final titrated daily dose established during the titration period.
  Other Names: FOSRENOL
  Arms: 1
Drug: Placebo — Placebo
  Arms: 2

SUMMARY:
Chronic kidney disease (CKD) can result in a loss of ability to filter and excrete phosphate. The body's attempt to adjust to an increased level of phosphate in the blood can result in elevated levels of hormones and minerals resulting in serious clinical consequences. This study is being conducted to evaluate the safety and efficacy of lanthanum carbonate in lowering high levels of phosphorus in the blood in subjects with CKD Stages 3 and 4 compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Under a physician's care for CKD for > 2 months and are not expected to begin dialysis for 4 months
* Screening estimated GFR of 15-59 mL/1.73 m2
* Serum phosphorus >= 4.7 mg/d following washout

Exclusion Criteria:

* Requiring treatment with cinacalcet HCI or compounds containing phosphate, aluminum, calcium or magnesium
* Rapidly progressing glomerulonephritis
* Cirrhosis or other clinically significant liver diseases
* Past or present uncontrolled peptic ulcer, Crohn's disease, malignancy or recent GI bleed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2006-01-11 (Actual); Primary Completion 2007-06-01 (Actual); Study Completion 2007-06-01 (Actual)

PRIMARY OUTCOMES:
Serum phosphorus levels at 8 weeks. | 8 weeks

SECONDARY OUTCOMES:
PTH levels, calcium-phosphorus product. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (10):
- United States (10):
  - VA Greater Los Angeles Health Care System, Los Angeles, California
  - Barnett Research & Communications Medical Corporation, Torrance, California
  - Western Nephrology & Metabolic Bone Disease, PC, Thornton, Colorado
  - Outcomes Research International, Inc., Hudson, Florida
  - Twin Cities Clinical Research, Brooklyn Center, Minnesota
  - St. Louis University/Nephrology, St Louis, Missouri
  - University of North Carolina, Chapel Hill, North Carolina
  - Northwest Renal Clinic, Portland, Oregon
  - Nephrology Associates, Nashville, Tennessee
  - Kidney Associates, Houston, Texas

REFERENCES:
- [Result] Sprague SM, Abboud H, Qiu P, Dauphin M, Zhang P, Finn W. Lanthanum carbonate reduces phosphorus burden in patients with CKD stages 3 and 4: a randomized trial. Clin J Am Soc Nephrol. 2009 Jan;4(1):178-85. doi: 10.2215/CJN.02830608. Epub 2008 Dec 3. PMID 19056618
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086
- See also: FDA Recall Information — http://www.fda.gov/opacom/7alerts.html